CLINICAL TRIAL: NCT00159042
Title: Identification of Novel Genetic Modifiers in Beta-thalassemia
Brief Title: Genetic Factors Affecting the Severity of Beta Thalassemia
Status: Completed | Type: Observational
Sponsor: Deborah Rund (Other)
Responsible Party: Sponsor-Investigator, Deborah Rund, Senior Hematologist, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: 302803-HMO-CTIL
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA isolated from peripheral blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with genetic diseases can have widely differing severities. We are looking for genetic factors which influence the severity of beta thalassemia.

DETAILED DESCRIPTION:
The understanding of the phenotypic variability of genetically homogeneous disorders represents a major challenge. In beta thalassemia, the beta globin gene is affected by a variety of mutations. The group of patients to be analyzed here is homozygous for a splice site mutation that is common in the Middle East. In contrast to this genetic homogeneity, the spectrum of the clinical phenotype ranges from mild anemia to most severe, transfusion dependent anemia. We will use a genetic linkage approach to identify modifying factors and by analyzing the efficiency of an mRNA surveillance mechanism that is referred to as nonsense-mediated decay and represents a candidate genetic modifier of beta thalassemia and other genetic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Identification of homozygous IVS1 nt 6 beta thalassemia mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients analyzed for beta thalassemia in our laboratory in Hadassah.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Oppenheim, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Rund D, Oron-Karni V, Filon D, Goldfarb A, Rachmilewitz E, Oppenheim A. Genetic analysis of beta-thalassemia intermedia in Israel: diversity of mechanisms and unpredictability of phenotype. Am J Hematol. 1997 Jan;54(1):16-22. doi: 10.1002/(sici)1096-8652(199701)54:13.0.co;2-7. PMID 8980256